CLINICAL TRIAL: NCT06257082
Title: Development of a Culturally Adapted, Video-based Patient Education Intervention to Increase Diabetic Eye Screening and Teleophthalmology Use in Latinx Communities
Brief Title: Video-based Patient Education Intervention for Diabetic Eye Screening in Latinx Communities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2024-1566; A536000 (Other: UW Madison); 1UG1EY032446-01 (NIH)
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Diabetic Retinopathy
Keywords: teleophthalmology
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Patient plus Clinician Combined Testimonials (Active Comparator): In addition to being randomized for online survey participants, focus groups will view patient plus clinician combined testimonials.
  Interventions: Other: Online Survey
- Clinician Only Testimonials (Active Comparator)
  Interventions: Other: Online Survey
- Patient Only Testimonials (Active Comparator)
  Interventions: Other: Online Survey
- National Eye Institute video Control (Active Comparator)
  Interventions: Other: Online Survey
- Pre-video questionnaire-only Control (Active Comparator)
  Interventions: Other: Online Survey

INTERVENTIONS:
Other: Online Survey — Participants must self-identify as Latinx adults and complete a brief online survey adapted from validated survey instruments for eye health literacy and trust in healthcare (CADEES and T-HCT scale) both before and after viewing the video-based, patient education intervention to obtain a pre to post-comparison of any differences in their responses.

SUMMARY:
An online survey (n=1,500) and 4 focus groups will be conducted with Latinx patients with diabetes (n=20) to obtain preliminary data regarding whether and how patient and clinician video testimonial interventions (n=6) increase eye health literacy and trust in healthcare.

DETAILED DESCRIPTION:
3 Latinx patients with diabetes and 3 Latinx clinicians will be recruited to videotape testimonials regarding the importance of diabetic eye screening and teleophthalmology use from their personal experiences. The investigators will structure the testimonials as a series of responses to a brief set of interview questions, or prompts, designed to elicit key messages previously identified by our community stakeholders as being particularly important, based on our prior studies and those of others and conducted in Spanish (with English subtitles).

After the Latinx patient and clinician video testimonials are recorded, a community outreach specialist bilingual in Spanish and English will facilitate a series of 4 community stakeholder meetings (90 min. each) to develop the culturally-adapted, video-based patient education intervention to increase diabetic eye screening and teleophthalmology use among Latinos.

After patient education videos are developed, an online survey will be conducted (n=1500) to test 3 versions of the video-based patient education intervention: (1) patient + clinician combined testimonials, (2) patient testimonials only, (3) clinician testimonials only, and compare them to 2 control conditions: (1) a standard educational video, publicly available online from the National Eye Institute, and (2) pre-video questionnaire-only control in a mixed-effects randomized design with pre- and post-measures (video conditions treated as the between-subjects factor).

Finally, a community outreach specialist bilingual in Spanish and English will facilitate focus groups (60-90 minutes) in the participants' preferred language (participants will be grouped based on their preference for either Spanish or English). Focus groups will begin by having each participant complete a brief survey instrument that will be read aloud and adapted from validated survey instruments for eye health literacy and trust in healthcare (CADEES and T-HCT scale). Participants will then silently view the video-based, patient education intervention (patient + clinician combined version). Afterwards, they will complete the same brief survey instrument to obtain a pre-/post-comparison of any differences in their responses that may result from viewing the video intervention.

Together with the online survey results, the investigators will test the intervention's ability to increase eye health literacy and trust in healthcare for obtaining eye care.

ELIGIBILITY:
Inclusion Criteria (online survey participants):

* Self-Identifies as Hispanic or Latino

Inclusion Criteria (patient video testimonials):

* Self-Identifies as Hispanic or Latino
* diagnosed with diabetes
* treated at Access Community Health Centers and UW Health in Madison, WI

Inclusion Criteria (clinician video testimonials):

* Self-Identifies as Hispanic or Latino
* clinician who treats patients with diabetes at Access Community Health Centers and UW Health in Madison, WI

Inclusion Criteria (focus group participants):

* Self-Identifies as Hispanic or Latino
* diagnosed with type 1 or type 2 diabetes

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1526 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in Eye Health Literacy as measured by Compliance with Annual Diabetic Eye Exams Survey (CADEES) | pre and post video testimonial intervention (up to 90 minutes)
  CADEES is scored from 1-5 where higher scores indicate increase eye health literacy.

SECONDARY OUTCOMES:
Change in Trust in Healthcare as measured by Trust in the Health Care Team (T-HCT) scale score | pre and post video testimonial intervention (up to 90 minutes)
  T-HCT is scored from 1-5 where higher scores indicate increased trust in healthcare.

CONTACTS AND LOCATIONS:
Overall Officials: Yao Liu, MD, MS, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- UW Hospital and Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data regarding patient demographics, whether they obtained diabetic eye screening, had teleophthalmology performed, any vision-threatening eye condition identified by teleophthalmology, and whether they followed-up for in-person eye care if they screened positive will be available to share.
Supporting Information: Study Protocol, SAP
Time Frame: up to 7 years after the completion of the primary outcome
Access Criteria: contact study PI for access

REFERENCES:
- See also: A Guide to Implementation for Sustained Impact in Teleophthalmology (I-SITE) — https://www.hipxchange.org/I-SITE
- See also: Implementation of Teleophthalmology in Urban Health Systems Study — https://clinicaltrials.gov/study/NCT05773495